CLINICAL TRIAL: NCT00959075
Title: A Randomized Controlled Trial of the Effect of Thiamin Supplementation on Heart Function in Ambulatory Patients With Heart Failure
Brief Title: A Trial of Thiamin Supplementation in Patients With Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA6617
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Heart Failure
Keywords: Thiamin supplementation; Thiamin deficiency; Heart failure; Improve heart function; Vitamin B1 supplementation
MeSH Terms: conditions — Heart Failure; Beriberi | interventions — Thiamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral thiamin supplementation (Experimental): Vitamin B1 (Oral thiamin) 100mg BID for 6 months
  Interventions: Dietary Supplement: Vitamin B1
- Sugar pill (Placebo Comparator): oral placebo 1 tablet BID for 6 months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin B1 — 100 mg Twice a day
  Other Names: Jamieson - Thiamin Mononitrate
  Arms: Oral thiamin supplementation
Dietary Supplement: Placebo — Sugar pill
  Arms: Sugar pill

SUMMARY:
Background: Patients with heart failure (HF) are at increased risk of developing thiamin deficiency (TD). Thiamin (vitamin B1) is required for the production of energy and therefore TD may contribute to the energy depletion commonly observed in the failing heart. Thiamin supplementation trials to date have shown conflicting results and therefore further studies to explain the impact of thiamin supplementation on HF patients with TD is necessary.

Objective: The purpose of this study is to determine whether thiamin supplementation in an ambulatory cohort of patients with systolic heart failure will provide any benefit in terms of improved heart function, symptoms, exercise capacity, and quality of life.

Description: Patients involved in the study will be given either thiamin supplements or a matching placebo (pills containing no thiamin) for 6 months. The ability of the heart to pump before and after the supplementation will be measured using cardiac magnetic resonance imaging (MRI)and/or 3D echocardiography.

Relevance: This study will determine whether thiamin supplementation improves cardiac function, exercise tolerance and quality of life. Thiamin supplementation is widely available, inexpensive, and safe. Therefore this trial may have a major impact on the optimal management of the expanding population of heart failure patients.

DETAILED DESCRIPTION:
Background: There is now accumulating evidence that patients with heart failure (HF) have a high prevalence of thiamin deficiency (TD). Since thiamin is a key cofactor in the enzyme systems that produce energy from both carbohydrates and fats, TD may contribute to the energy depletion frequently observed in the failing heart. Altered energy reserves with a reduction in myocardial ATP have now been recognized to play a critical role in the development and progression of HF. Therefore, correction of TD may enhance cardiac energy substrate availability and utilization, leading to improvement of ventricular function and symptoms.

Primary Hypothesis: The left ventricular ejection fraction in stable, ambulatory patients with systolic heart failure receiving 6 months of oral thiamin supplementation will be significantly higher in comparison with those receiving a placebo.

Secondary Hypothesis: In heart failure patients oral thiamin supplementation will 1)have favourable effects on ventricular remodelling (reduction in diastolic and systolic volumes) and regional function; 2)reduce neurohormonal stimulation (BNP and norepinephrine) as well as oxidative stress; 3)improve exercise capacity and 4)improve symptoms and quality of life.

Ambulatory patients attending heart failure clinics at Mount Sinai, University Health Network, Trillium Health Centre and St. Michael's Hospital with systolic heart failure (NYHA class II-IV, left ventricular ejection fraction <45%) will be screened for eligibility to participate in our randomized trial. We will randomize seventy eligible patients using a stratified, permuted block randomization scheme, to be given either 100mg BID of thiamin HCl or a matching placebo BID in a 1:1 ratio to be taken for six months. All study personnel will be blinded to treatment assignment.

Participants will have baseline and follow-up visits which include collecting demographic data, history of medication use, symptoms, anthropometrics as well as a physical exam. Left ventricular ejection fraction, volumes, and regional function will be measured using a standardized echocardiogram and cardiac MRI at baseline and after six months of supplementation. At this time, blood markers of thiamin status, oxidative stress (F2 isoprostanes) and neurohormonal activation (norepinephrine and BNP) will also be measured. Participants will also complete a six-minute walk test, a 3-day dietary record, the Living with Heart Failure quality of life instrument and a 24-hour urine collection (to measure urinary thiamin excretion) at both baseline and follow-up visits. Compliance will be measured using returned pill counts and verified by measuring plasma thiamin levels which respond rapidly to thiamin supplementation.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of ischemic, dilated, idiopathic or valvular heart failure characterized by an ejection fraction of < 45% (echocardiography or radionuclide scan)
* have an optimized medication regimen (ACE inhibitor or angiotensin receptor blocker, and beta blocker at target doses, or up-titrated to the maximum doses as tolerated)
* been stable (on current medication regimen with no hospitalizations for acute decompensated heart failure > 2 months) prior to entry into the study

Exclusion Criteria: Participants will be excluded if they are:

* unable or unwilling to provide informed consent
* have any concurrent condition which would result in thiamin deficiency, namely gastrointestinal disorders, magnesium deficiency, liver disease, thyrotoxicosis, B12 deficiency, folate deficiency, prolonged diarrhoeal disease, dialysis, prolonged fever or infection, recent myocardial infarction, coronary revascularization (percutaneous coronary intervention or coronary artery bypass surgery within 3 months), or renal failure
* are rapidly deteriorating, who are not on a stable medication regimen (2 months or more) or who have been hospitalized for acute decompensated heart failure in the last 2 months
* are on experimental medications
* are taking vitamin supplements containing thiamin >10mg/day
* consume excessive alcohol (> 3 drinks per day), have a documented history of alcoholism or have documented alcoholic cardiomyopathy
* have permanent atrial fibrillation
* are pregnant or would like to become pregnant
* have a right-to-left, bidirectional, or transient right to left cardiac shunts
* have clinically suspected wet Beri Beri in the opinion of the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction measured by CMR or 3D echo at 6 months | 6 months

SECONDARY OUTCOMES:
LV volume, regional function as measure by CMR tagging | 6 months
Exercise tolerance - distance walked in the standard six-minute walk test | 6 months
Levels of circulating BNP, norepinephrine and F2-isoprostanes | 6 months
Scores on the Living with Heart Failure quality of life instrument | 6 months
Prevalence of TD in an ambulatory HF population | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary E. Keith, PhD, RD, Principal Investigator — Unity Health Toronto
Locations (1):
- Niagara North Family Health Team, St. Catharines, Ontario, Canada

REFERENCES:
- [Derived] Keith M, Quach S, Ahmed M, Azizi-Namini P, Al-Hesayen A, Azevedo E, James R, Leong-Poi H, Ong G, Desjardins S, Lee PJ, Ravamehr-Lake D, Yan AT. Thiamin supplementation does not improve left ventricular ejection fraction in ambulatory heart failure patients: a randomized controlled trial. Am J Clin Nutr. 2019 Dec 1;110(6):1287-1295. doi: 10.1093/ajcn/nqz192. PMID 31504093